CLINICAL TRIAL: NCT03431818
Title: Effective Fraction of Inspired Oxygen in Premature Infants Receiving Support Via Nasal Cannula
Brief Title: Effective Fraction of Inspired Oxygen With Nasal Cannula in Premature Infants
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nelson Claure, Associate Professor, University of Miami
Other Study IDs: 20170816
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Oxygen Therapy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nasal cannula flow rate — This is a crossover study where observations will be obtained at five nasal cannula flow rates: 0.5, 1, 2, 4 and 6 liters per minute.

SUMMARY:
The objective of this study is to determine the multifactorial relationship between the effective fraction of inspired oxygen (Effective-FiO2) and the FiO2 in the gas delivered by the nasal cannula (NC-FiO2), NC flow rate, spontaneous minute ventilation and other patient characteristics in premature infants who receive supplemental oxygen via nasal cannula (NC).

DETAILED DESCRIPTION:
During routine nasal cannula (NC) use in the newborn ICU, the actual fraction of oxygen inspired by the infant, i.e. the effective FiO2 (Effective-FiO2) that reaches the infant's airways, cannot be easily determined. The effective FiO2 during NC use is generally lower than the FiO2 in the gas delivered by NC at the infant's nose due to dilution with ambient gas entrained by the infants during spontaneous inspiration. The factors influencing effective FiO2 include the set FiO2 of the gas delivered by NC (NC-FiO2), the NC-flow rate, and the entrainment of ambient gas by the infant during each spontaneous inspiration. The individual contribution of each of these factors to the variability in effective-FiO2 in extreme premature infants has not been systematically evaluated.

The objective of this study is to determine the multifactorial relationship between the effective fraction of inspired oxygen (Effective-FiO2) and the FiO2 in the gas delivered by the nasal cannula (NC-FiO2), NC flow rate, spontaneous minute ventilation and other patient characteristics in premature infants who receive supplemental oxygen via nasal cannula (NC).

ELIGIBILITY:
Inclusion Criteria:

* Premature infants born between 23 and 30 weeks of gestational age
* Receiving supplemental oxygen via nasal cannula
* Parental informed consent

Exclusion Criteria:

* Major congenital anomalies
* Clinically unstable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature infants admitted to the newborn ICU will be screened. Infants who meet the inclusion criteria will be enrolled in the study after written informed parental consent is obtained:
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Nasal cannula FiO2 | from birth upto 40 weeks corrected postmenstrual age
  FiO2 necessary to maintain the effective FiO2 (measured at the hypopharynx) at the basal level at different nasal cannula flow rates.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Claure, Principal Investigator — University of Miami; Eduardo Bancalari, Principal Investigator — University of Miami; Deepak Jain, Principal Investigator — University of Miami
Locations (1):
- NICU at Holtz Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No